CLINICAL TRIAL: NCT02228889
Title: Prospective Trial Comparing the Performance Profiles of Two Non-Cross-Linked Porcine Dermal Matrices in Abdominal Wall Reconstruction
Brief Title: RCT of Two Noncrosslinked Porcine Acellular Dermal Matrices in Ab Wall Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeffrey Janis (Other)
Responsible Party: Sponsor-Investigator, Jeffrey Janis, Professor of Plastic Surgery, Vice-Chairman, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014H0041
Record Dates: First submitted 2014-08-18; First posted 2014-08-29 (Estimated); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Hernia, Ventral; Intestinal Fistula; Fibromatosis, Abdominal
Keywords: Hernia; Abdominal wall reconstruction; Abdominal wall defect; Porcine mesh; Component separation; Abdominal wall tumor; Desmoid
MeSH Terms: conditions — Hernia, Ventral; Intestinal Fistula; Fibromatosis, Abdominal; Hernia; Peritoneal Neoplasms; Desmoid Tumors | interventions — Abdominoplasty; strattice

STUDY DESIGN:
Intervention Model Description: Abdominal wall reconstruction using Strattice
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strattice (Experimental): Abdominal wall reconstruction with Strattice Assess pain intensity at last office visit preoperatively Assess pain interference at last office visit preoperatively Assess physical functioning at last office visit preoperatively Assess patient quality of life at last office visit preoperatively Assess patient pain intensity postoperatively Assess pain interference postoperatively Assess physical functioning postoperatively Assess quality of life postoperatively Assess hernia recurrence at 30 days postoperatively Assess bulge at 30 days postoperatively Assess Surgical Site Occurrences at 30 days postoperatively Assess hernia recurrence at 1 year postoperatively Assess bulge at 1 year postoperatively Assess Surgical Site Occurrences at 1 year postoperatively Assess overall complications at 30 days postoperatively Assess overall complications at 1 year postoperatively
  Interventions: Procedure: Abdominal wall reconstruction with Strattice; Other: Assess pain intensity at last office visit preoperatively; Other: Assess pain interference at last office visit preoperatively; Other: Assess physical functioning at last office visit preoperatively; Other: Assess patient quality of life at last office visit preoperatively; Other: Assess patient pain intensity postoperatively; Other: Assess pain interference postoperatively; Other: Assess physical functioning postoperatively; Other: Assess quality of life postoperatively; Other: Assess hernia recurrence at 30 days postoperatively; Other: Assess bulge at 30 days postoperatively; Other: Assess Surgical Site Occurrences at 30 days postoperatively; Other: Assess hernia recurrence at 1 year postoperatively; Other: Assess bulge at 1 year postoperatively; Other: Assess Surgical Site Occurrences at 1 year postoperatively; Other: Assess overall complications at 30 days postoperatively; Other: Assess overall complications at 1 year postoperatively; Device: Strattice
- XenMatrix (Experimental): Abdominal wall reconstruction with XenMatrix Assess pain intensity at last office visit preoperatively Assess pain interference at last office visit preoperatively Assess physical functioning at last office visit preoperatively Assess patient quality of life at last office visit preoperatively Assess patient pain intensity postoperatively Assess pain interference postoperatively Assess physical functioning postoperatively Assess quality of life postoperatively Assess hernia recurrence at 30 days postoperatively Assess bulge at 30 days postoperatively Assess Surgical Site Occurrences at 30 days postoperatively Assess hernia recurrence at 1 year postoperatively Assess bulge at 1 year postoperatively Assess Surgical Site Occurrences at 1 year postoperatively Assess overall complications at 30 days postoperatively Assess overall complications at 1 year postoperatively
  Interventions: Other: Assess pain intensity at last office visit preoperatively; Other: Assess pain interference at last office visit preoperatively; Other: Assess physical functioning at last office visit preoperatively; Other: Assess patient quality of life at last office visit preoperatively; Other: Assess patient pain intensity postoperatively; Other: Assess pain interference postoperatively; Other: Assess physical functioning postoperatively; Other: Assess quality of life postoperatively; Other: Assess hernia recurrence at 30 days postoperatively; Other: Assess bulge at 30 days postoperatively; Other: Assess Surgical Site Occurrences at 30 days postoperatively; Other: Assess hernia recurrence at 1 year postoperatively; Other: Assess bulge at 1 year postoperatively; Other: Assess Surgical Site Occurrences at 1 year postoperatively; Other: Assess overall complications at 30 days postoperatively; Other: Assess overall complications at 1 year postoperatively; Procedure: Abdominal wall reconstruction with XenMatrix; Device: XenMatrix

INTERVENTIONS:
Procedure: Abdominal wall reconstruction with Strattice — Abdominal wall reconstruction using Strattice
  Arms: Strattice
Other: Assess pain intensity at last office visit preoperatively — Assess patient pain intensity preoperatively using the PROMIS Pain Intensity survey (average of 1-3 weeks preoperatively)
Other: Assess pain interference at last office visit preoperatively — Assess pain interference preoperatively using the PROMIS pain interference survey (average of 1-3 weeks preoperatively)
Other: Assess physical functioning at last office visit preoperatively — Assess physical functioning preoperatively using the PROMIS physical functioning survey (average of 1-3 weeks preoperatively)
Other: Assess patient quality of life at last office visit preoperatively — Assess patient quality of life preoperatively, using the HerQLes survey (average of 1-3 weeks preoperatively)
Other: Assess patient pain intensity postoperatively — Assess patient pain intensity at 1 year postoperatively using the PROMIS Pain Intensity survey
Other: Assess pain interference postoperatively — Assess pain interference at 1 year postoperatively using the PROMIS Pain Interference survey
Other: Assess physical functioning postoperatively — Assess physical functioning at 1 year postoperatively using the PROMIS Physical Functioning Survey
Other: Assess quality of life postoperatively — Assess quality of life at 1 year postoperatively using the HerQLes survey
Other: Assess hernia recurrence at 30 days postoperatively — Assess hernia recurrence at 30 days
Other: Assess bulge at 30 days postoperatively — Assess bulge at 30 days
Other: Assess Surgical Site Occurrences at 30 days postoperatively — Assess Surgical Site Occurrences at 30 days
Other: Assess hernia recurrence at 1 year postoperatively — Assess hernia recurrence at 1 year postoperatively
Other: Assess bulge at 1 year postoperatively — Assess bulge at 1 year postoperatively
Other: Assess Surgical Site Occurrences at 1 year postoperatively — Assess Surgical Site Occurrences at 1 year postoperatively
Other: Assess overall complications at 30 days postoperatively
Other: Assess overall complications at 1 year postoperatively
Procedure: Abdominal wall reconstruction with XenMatrix — Abdominal wall reconstruction with XenMatrix
  Arms: XenMatrix
Device: Strattice — Strattice mesh
  Arms: Strattice
Device: XenMatrix — Xenmatrix mesh
  Arms: XenMatrix

SUMMARY:
The purpose of the study is to compare the clinical outcomes of two commonly used, FDA-approved biologic meshes in hernia repair and abdominal wall reconstruction (Strattice and XenMatrix). The two meshes are derived from pig skin from which cells have been removed and which have been sterilized. The two meshes are made by two different companies using different processes.

DETAILED DESCRIPTION:
This is a prospective, randomized-controlled trial comparing two porcine acellular matrices in abdominal wall reconstruction. It is single-blind (patients are blinded to the type of mesh used while surgeons are not).

Our goals in this study are:

1. PRIMARY OUTCOME: To compare the overall complication rates between two non-cross-linked porcine dermal matrices (XenMatrix and Strattice) at 30 days and 1 year postoperatively
2. SECONDARY OUTCOMES

i. To compare the rate of Surgical Site Occurrences (SSOs) between XenMatrix and Strattice in abdominal wall reconstruction at 30 days and 1 year postoperatively

1. Infection
2. Seroma
3. Hematoma
4. Wound dehiscence
5. Skin necrosis
6. Formation of enterocutaneous fistula
7. Mesh infection ii. To compare the hernia recurrence rate between XenMatrix and Strattice at 30 days and 1 year postoperatively iii. To compare the bulge rate between XenMatrix and Strattice at 30 days and 1 year postoperatively iv. To compare to changes in patient pain, physical functioning and quality of life after hernia repair between XenMatrix and Strattice, preoperatively, and at 1 year postoperatively A. Pain assessment: Patient Reported Outcomes Measurement Information System (PROMIS) Pain Intensity survey, PROMIS Pain Interference survey B. Physical functioning assessment: PROMIS Physical Function C. Quality of life assessment: Hernia-Related Quality-of-Life (HerQLes) survey

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Patients presenting for elective hernia repair, with Ventral Hernia Working Group (VHWG) grade 2 or above (Patients with a hernia who need hernia repair due to hernia size, discomfort, risk of bowel incarceration, effect on physical function), and who have comorbidities or contamination making the use of synthetic mesh contraindicated)
* Patients deemed to be good surgical candidates, with no active life-threatening cardiac disease, pulmonary disease, renal disease, hematologic disease (patients who can have a major surgical procedure without an exceedingly high risk of medical complications such as pulmonary edema, myocardial infarction, pulmonary embolism, renal failure, life-threatening bleeding, stroke).
* Patients presenting for resection of large abdominal wall tumors who are expected to undergo have tumor extirpative defect that would require biologic mesh for closure (patients with a large tumor of the abdominal wall who will have a large defect in their fascia after resection, who need biologic mesh for reinforcement).

Exclusion Criteria:

* Known allergy to porcine products
* Active smokers (within the past 4 weeks) presenting for elective hernia repair
* Patients with active life-threatening cardiac disease, pulmonary disease, renal disease, hematologic disease presenting for elective hernia repair
* Patients presenting for emergent hernia repair (in the setting of bowel strangulation, necrosis, penetrating trauma) as it will be difficult to consent those patients for the study preoperatively
* Patients with severe systemic sepsis
* Patients with frank purulence in the wound

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey E Janis, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were no significant events in the study. Enrollment was stopped prior to the pre-determined 70 total participants, as a shift in practice and national trend toward the use of synthetic mesh over biologic mesh hindered participant recruitment.
Groups:
- Strattice: Abdominal wall reconstruction with Strattice Assess hernia recurrence at 30 days postoperatively Assess bulge at 30 days postoperatively Assess Surgical Site Occurrences at 30 days postoperatively Assess hernia recurrence at 1 year postoperatively Assess bulge at 1 year postoperatively Assess Surgical Site Occurrences at 1 year postoperatively Assess overall complications at 30 days postoperatively Assess overall complications at 1 year postoperatively
- XenMatrix: Abdominal wall reconstruction with XenMatrix Assess hernia recurrence at 30 days postoperatively Assess bulge at 30 days postoperatively Assess Surgical Site Occurrences at 30 days postoperatively Assess hernia recurrence at 1 year postoperatively Assess bulge at 1 year postoperatively Assess Surgical Site Occurrences at 1 year postoperatively Assess overall complications at 30 days postoperatively Assess overall complications at 1 year postoperatively
Period: Overall Study
Arm/Group | Strattice | XenMatrix
Started | 16 | 30
Completed | 16 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrollment was stopped prior to the pre-determined 70 total participants, as a shift in practice and national trend toward the use of synthetic mesh over biologic mesh hindered participant recruitment.
Groups:
- Strattice; XenMatrix: Assess Bulge Assess Surgical Site Occurrences at 6 weeks Assess Recurrence Assess Seroma Assess Hematoma Assess Infection Assess Dehiscence Assess Skin necrosis
- Total: Total of all reporting groups
Arm/Group | Strattice | XenMatrix | Total
Number analyzed (Participants) | 16 | 30 | 46
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [55.8 to 68.6] | 57 [43 to 62.1] | 60 [43 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 6 | 16 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 29.6 [26.8 to 33.5] | 33.1 [26.5 to 37.4] | 33.1 [26.4 to 37.3]
Number of prior Hernia Repairs [Median (Inter-Quartile Range); unit: prior repairs] | 2.5 [0 to 9] | 1 [0 to 2] | 1 [0 to 4.5]
Hernia Width [Median (Inter-Quartile Range); unit: cm] | 15.8 [10 to 18.7] | 12.9 [9.5 to 18.7] | 12.9 [9.48 to 18.71]
Diabetes [Count of Participants; unit: Participants] | 7 | 7 | 14
Hypertension [Count of Participants; unit: Participants] | 7 | 14 | 21
COPD [Count of Participants; unit: Participants] | 5 | 5 | 10
Immunosuppression [Count of Participants; unit: Participants] | 2 | 10 | 12
Previous Hernia Repair [Count of Participants; unit: Participants] | 11 | 20 | 31
ASA Class [Count of Participants; unit: Participants] — Participants are clinically graded using the ASA Physical Status Classification System, based on their overall health status and systemic disease burden at the time of surgery. Lower grades correlate to better outcomes. Stages I-II are better outcomes with Stages III-V are worse outcomes. lower ASA classes (I-II) are associated with better surgical outcomes, while higher classes (III-V) indicate increased risk of complications. This staging reflects overall health and is used both clinically and in research to stratify risk.
  Participants
    Stage I | 0 | 0 | 0
    Stage II | 3 | 3 | 6
    Stage IIII | 13 | 24 | 37
    Stage IV | 0 | 3 | 3
    Stage V | 0 | 0 | 0
Ventral Hernia Working Group [Count of Participants; unit: Participants] — VHWG grading system categorizes patients based on the risk of surgical site occurrences (SSOs) and wound complications during ventral hernia repair. It incorporates host comorbidities, wound condition, and presence of infection. Grades 1-2 correlate with better outcomes, Grades 3-4 are worse outcomes. VHWG Grades 1-2 are associated with favorable surgical outcomes, while Grades 3-4 represent higher-risk patients with significantly increased complication rates due to infection or contamination.
  Participants
    1 | 1 | 1 | 2
    2 | 2 | 9 | 11
    3 | 11 | 13 | 24
    4 | 2 | 7 | 9
Kanters Grade [Count of Participants; unit: Participants] — Kanters Grade categorizes patients based on the severity and complexity of the hernia and overall health. This helps predict the risk of complications, wound infections and hernia recurrence. Grade 1-2 are correlated with better outcomes and Grade 3-4 are worse outcomes. Grades 1 and 2 are associated with better outcomes, such as lower complication rates, quicker recovery, and the ability to use synthetic mesh. Kanters Grades 3 and 4 represent more complex hernias with higher complication risks, including infection, need for biologic mesh, longer recovery times, and higher recurrence rates
  Participants
    1 | 1 | 1 | 2
    2 | 6 | 16 | 22
    3 | 9 | 13 | 22
Primary Fascial Repair [Count of Participants; unit: Participants] | 14 | 22 | 36
Unilateral Component Separation [Count of Participants; unit: Participants] | 2 | 2 | 4
Bridged Repair [Count of Participants; unit: Participants] | 2 | 6 | 8
Total OR Time [Median (Inter-Quartile Range); unit: minutes] | 471 [444 to 484] | 417 [336 to 548] | 417 [336 to 547]

OUTCOME MEASURES:

1. Primary Outcome: Rate of Surgical Site Occurrences (SSOs) at 6 Week
Description: Compare the rate of Surgical Site Occurrences (SSOs) between XenMatrix and Strattice in abdominal wall reconstruction at 1 year postoperatively. These include:
  1. Infection
  2. Seroma
  3. Hematoma
  4. Wound dehiscence
  5. Skin necrosis
  6. Formation of enterocutaneous fistula
  7. Mesh infection
Time Frame: 6 week postoperatively
Population: participants who got to 6 weeks
Measure: Mean (Standard Error); unit: event
Arm/Group | Strattice | XenMatrix
Number analyzed (Participants) | 16 | 30
event | 1 (6.25) | 11 (36.67)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Strattice: Infections: Infections at the surgical site or throughout the body are a potential risk.
  Seromas: Fluid collections (seromas) can form at the surgical site. Wound Healing Problems: Necrosis (tissue death) or impaired wound healing can occur.
  Wound Dehiscence: The wound may reopen. Implant Exposure: In some cases, the breast implant may become exposed. Hematoma: Blood clots can form at the surgical site. Erythema: Redness or inflammation of the skin. Explantation: In some cases, the implant may need to be removed (explanted). Re-implantation of an expander: In some cases, a breast expander may need to be re-implanted.
  Salvage procedures: In some cases, additional procedures may be needed to address complications.
  Implant Loss: In rare cases, the implant may be lost.
- XenMatrix: Allergic Reactions: Hypersensitivity to porcine products or tetracyclines/rifamycins is a contraindication for using XenMatrix.
  Seroma: A collection of fluid under the skin or tissue. Infection: The surgical site or the graft itself can become infected. Inflammation: Swelling and redness around the surgical area. Adhesion: Scar tissue forming between tissues or organs. Fistula formation: An abnormal connection or passage between two organs or tissues.
  Erosion: Wearing away or breakdown of the tissue. Hematoma: A collection of blood outside of a blood vessel. Recurrence of the tissue defect: The hernia or tissue defect returns after surgery.
  Wound Dehiscence: The wound opening up after surgery. Hernia Recurrence: The hernia returns after surgery.
Arm/Group | Strattice | XenMatrix
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/30
Other Adverse Events (participants affected / at risk) | 0/16 | 0/30

LIMITATIONS AND CAVEATS:
The study was completed prior to the anticipated 70 total participants, as new data and literature have shifted a national trend away from the use of biologic mesh and toward synthetic mesh, which significantly impeded recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2024-09-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT02228889/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-18): https://cdn.clinicaltrials.gov/large-docs/89/NCT02228889/SAP_001.pdf
  • Informed Consent Form (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT02228889/ICF_002.pdf